CLINICAL TRIAL: NCT06088472
Title: A Single-arm Phase I Clinical Study of TIL Injection for the Treatment of Metastatic or Recurrent Solid Tumors
Brief Title: TIL Injection for the Treatment of Metastatic or Recurrent Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CO-FA-012
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumors, Adult
MeSH Terms: interventions — Toll-Like Receptor 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TIL injection treatment group (Experimental)
  Interventions: Biological: TIL injection

INTERVENTIONS:
Biological: TIL injection — Autologous tumor infiltrating lymphocyte injection

SUMMARY:
This is a single-center, single-arm phase I clinical trial.The study process was divided into: screening period, sampling and production period, NMA-LD chemotherapy , treatment and observation period, and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in the study, sign the informed consent form, and be willing and able to follow the study protocol ;
* 2.Must have a confirmed diagnosis of malignancy of their receptive histologies or cytologies: unresectable recurrent or metastatic solid tumor;
* 3.At least one resectable lesion (preferably superficial metastatic lymph nodes) that has not been treated with radiation and has not received other local therapies, and at least tissue blocks with a volume of≥0.5 cubic centimeter (either of single lesion origin or multiple lesions combined) can be isolated for the preparation of autologous tumor-infiltrating lymphocytes. Minimally invasive treatment where possible;

Exclusion Criteria:

* 1. Patients who have symptomatic and/or untreated CNS metastases (Except stable brain metastases, no medication required within 3 months, no hormone dependence);
* 2.The patient who has any active autoimmune disease, history of autoimmune disease, need for systemic steroid hormones or a condition requiring immunosuppressive drug therapy (>10 mg/day of prednisone or equivalent hormone) within 14 days before lymphocyte depletion chemotherapy;
* 3. Arterial/venous thrombotic events within 6 months prior to enrollment, such as: cerebrovascular accident, deep vein thrombosis and pulmonary embolism occurring;
* 4.Active infections requiring treatment with systemic anti-infectives (except for topical antibiotics); or those with unexplained fever > 38.5℃ occurring during the screening period, except for tumor fever;
* 5. Patients who have refractory or intractable epilepsy, hydrops abdominis, active gastrointestinal bleeding or IL-2 contraindications;
* 6. Patients who have received allogeneic bone marrow transplantation or an organ allograft;
* 7.Patients who have a history of hypersensitivity to any component or excipient of study drugs: autologous tumor infiltrating lymphocytes, cyclophosphamide, fludarabine, IL-2, dimethyl sulfoxide (DMSO), human serum albumin (HSA), dextran-40 and antibiotics (beta lactam antibiotics, gentamicin);

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events per CTCAE 5.0 | From TIL infusion to the 24th week
  To characterize the safety profile of autologous TIL injection (GT101) in patients with relapsed/metastatic advanced solid tumor as measured by the incidence and severity of adverse events per CTCAE 5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 24 months post infusion
  To evaluate the proportion of participants who have a confirmed partial response (PR) and complete response (CR) per RECIST v1.1 and iRECIST as assessed by the investigator.
Disease control rate (DCR) | Up to 24 months post infusion
  To evaluate the percentage of participants that achieved partial response (PR), complete response (CR), or stable disease (SD) after treatment among total number of evaluable patients.
Progression-free survival (PFS) | Up to 24 months post infusion
  To evaluate the time from the date of TIL infusion until disease progression per RECIST v1.1 and iRECIST as assessed by the investigator or death due to any cause.
Duration of Response (DoR) | Up to 24 months post infusion
  To evaluate the duration from the time that criteria are met for CR or PR per RECIST v1.1 and iRECIST as assessed by the investigator until disease progression or death due to any cause.
Overall survival (OS) | From the date of TIL infusion to date of death due to any cause, or up to 24 months post infusion (whichever occurs first)
  To evaluate the time from the date of TIL infusion to death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No